CLINICAL TRIAL: NCT05882045
Title: A Randomized, Double-Blind, Phase 3 Study to Investigate the Efficacy and Safety of LY3437943 Once Weekly Compared to Placebo in Participants With Severe Obesity and Established Cardiovascular Disease
Brief Title: A Study of Retatrutide (LY3437943) in Participants With Obesity and Cardiovascular Disease
Acronym: TRIUMPH-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18582; J1I-MC-GZBM (Other: Eli Lilly and Company); 2023-503659-88-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of retatrutide once weekly in participants with obesity and established cardiovascular disease (CVD). The study will last about 113 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥35.0 kilogram/square meter (kg/m²).
* Have established cardiovascular (CV) disease with at least 1 of the following:

  * prior myocardial infarction
  * prior ischemic or hemorrhagic stroke, or
  * symptomatic peripheral arterial disease
* Have a history of at least 1 self-reported unsuccessful dietary effort to reduce body weight.

Exclusion Criteria:

* Have had acute myocardial infarction, stroke, coronary revascularization, hospitalization for unstable angina, or hospitalization due to congestive heart failure within 90 days prior to screening.
* Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
* Have a prior or planned surgical treatment of obesity.
* Have a change in body weight greater than 5 kg (11 pounds) within 90 days prior to screening.
* Have Type 1 diabetes.
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 80

SECONDARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 80
Change from Baseline in Waist Circumference | Baseline, Week 80
Percent Change from Baseline in Total Cholesterol | Baseline, Week 80
Percent Change from Baseline in Triglycerides | Baseline, Week 80
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 80
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 80
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 80
Percent Change from Baseline in Fasting Insulin | Baseline, Week 80
Change from Baseline in Short Form version 2 (SF-36v2) Acute Form Physical Function Domain Score | Baseline, Week 80
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Cure (AUC) | Baseline to Week 80
  AUC is presented as a single average measure of AUC across the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (169):
- United States (46):
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Valley Clinical Trials, Inc., Covina, California
  - Neuro-Pain Medical Center, Fresno, California
  - Valley Research, Fresno, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Velocity Clinical Research, Panorama City, Van Nuys, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Humphreys Diabetes Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Great Lakes Clinical Trials - Gurnee, Gurnee, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Brengle Family Medicine, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - MedVadis Research Corporation, Waltham, Massachusetts
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - UPMC Montefiore University Hospital, Pittsburgh, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Tribe Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Advanced Research Institute, Ogden, Utah
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (24):
  - CEDIC, CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires, Buenos Aires
  - MICA - Medicina e Investigación Cardiometabólica, Del Viso, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - Stat Research S.A., Buenos Aires, Buenos Aires F.D.
  - Investigaciones Medicas Imoba Srl, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Centro Medico Privado San Vicente Diabetes, Córdoba, Córdoba Province
  - Centro de Salud e Investigaciones Médicas, Santa Rosa, La Pampa Province
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria, Santa Fe Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Fundación Respirar, Buenos Aires
  - Instituto Médico DAMIC, Córdoba
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Sanatorio Norte, Santiago del Estero
- Australia (19):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Emeritus Research, Botany, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Camden Hospital, Camden, New South Wales
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - University of Sydney - Charles Perkins Centre, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Core Research Group, Brisbane, Queensland
  - CDH Research Institute, Maroochydore, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Fusion Clinical Research, Adelaide, South Australia
  - Nightingale Research, Adelaide, South Australia
  - Southern Adelaide Diabetes & Endocrine Services, Mount Gambier, South Australia
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg West, Victoria
  - One Clinical Research, Nedlands, Western Australia
- Canada (17):
  - BC Diabetes Office, Vancouver, British Columbia
  - Discovery Clinical Services, Victoria, British Columbia
  - Joanne F. Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - Dr. Steven V. Zizzo Research Professional Corporation, Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Centricity Research Oshawa, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Manna Research Toronto, Toronto, Ontario
  - Ecogene-21 - Cmas, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique de médecine Urbaine du Quartier Latin, Montreal, Quebec
  - CardioVasc HR Inc, Saint-Jean-sur-Richelieu, Quebec
  - Centre de Medecine Metabolique de Lanaudiere (CMML), Terrebonne, Quebec
  - C.I.C. Mauricie inc., Trois-Rivières, Quebec
  - Syneos Health, Québec
- Hungary (12):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Regia Med Kft, Székesfehérvár, Fejér
  - Medifarma 98 Kft, Nyíregyháza, Nyíregyháza
  - Szent Lázár Megyei Kórház, Salgótarján, Nógrád megye
  - Óbudai Egészségügyi Centrum - Kaposvár Site, Kaposvár, Somogy County
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg, Zala County
  - Óbudai Egészségügyi Centrum, Budapest
  - ClinDiab Kft., Budapest
  - TRANTOR'99 Bt. Anyagcsere Centrum, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Óbudai Egészségügyi Centrum - Zalaegerszeg, Zalaegerszeg
- Mexico (16):
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana, Estado de Baja California
  - Centro Multidisciplinario de Diabetes de Pachuca, Pachuca, Hidalgo
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C., Zapopan, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - IMED Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Eukarya PharmaSite, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - EME RED Hospitalaria, Mérida, Yucatán
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Investigacion En Salud Y Metabolismo S.C / Nutricion Clinica / Unidad de Base de Datos, Chihuahua City
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Centro de Atención e Investigación Cardiovascular del Potosí, San Luis Potosí City
  - FAICIC S. de R.L. de C.V., Veracruz
- Poland (9):
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - NBR Polska, Warsaw, Masovian Voivodeship
  - KLIMED Marek Klimkiewicz, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - NZOZ Salvia CM, Katowice, Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 SUM, Zabrze, Silesian Voivodeship
  - Ambulatorium Sp. z o.o., Elblag, Warmian-Masurian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Puerto Rico (3):
  - Ponce Medical School Foundation Inc., Ponce
  - Clinical Research Management Group Inc, Ponce
  - Latin Clinical Trial Center, San Juan
- Slovakia (9):
  - Nemocnica s poliklinikou Lucenec, Lučenec, Banská Bystrica Region
  - Metabol KLINIK, Bratislava, Bratislava Region
  - MediVet s.r.o., Malacky, Bratislava Region
  - Human Care s.r.o., Košice, Košice Region
  - Tatratrial s.r.o., Rožňava, Košice Region
  - Areteus s.r.o., Trebišov, Košice Region
  - MEDI-DIA s.r.o., Sabinov, Presov
  - MediTask, Bratislava
  - Diab - Int, Bytča, Žilina Region
- Spain (14):
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol, A Coruña [La Coruña]
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Hospital Universitari Son Espases, Palma, Balears [Baleares]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Virgen del Camino, Sanlúcar de Barrameda, Cádiz
  - Hospital Virgen de las Montañas, Villamartín, Cádiz
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [Lérida]
  - Vithas Hospital Sevilla, Seville, Sevilla
  - Hospital Universitario de La Ribera, Alzira, Valenciana, Comunitat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants With Obesity and Cardiovascular Disease (TRIUMPH-3) — https://trials.lilly.com/en-US/trial/405675